CLINICAL TRIAL: NCT02842463
Title: Use of the 6-minute Stepper Test to Individualise Pulmonary Rehabilitation in Patients With Mild to Moderate Chronicle Obstructive Pulmonary Disease
Brief Title: 6-minute Stepper Test and Pulmonary Rehabilitation in Patients With Chronicle Obstructive Pulmonary Disease
Acronym: 6STaR
Status: Completed | Type: Observational
Sponsor: ADIR Association (Other)
Responsible Party: Sponsor
Other Study IDs: 6STaR
Record Dates: First submitted 2016-07-19; First posted 2016-07-25 (Estimated); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Pulmonary Rehabilitation; 6-minute Stepper Test
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Prospective observational cohort: Every patient referred to pulmonary rehabilitation program will be eligible. They will perform cardiopulmonary exercise testing prior to join rehabilitation program.
  During the first session of pulmonary rehabilitation, they will perform 2 6-minute stepper test with a rest of 20 minutes minimum between each test.
  Interventions: Other: 2 times : 6-minute stepper test with a rest of 20min between each test.

INTERVENTIONS:
Other: 2 times : 6-minute stepper test with a rest of 20min between each test.

SUMMARY:
The purpose of this study is to determine, if it exists, a relation between plateau heart rate from the last 3 minutes of the 6-minute stepper test and heart rate from first ventilatory threshold from cardiopulmonary exercise testing in order to individualise pulmonary rehabilitation in patients with mild to moderate chronicle obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 ans ;
* Chronicle obstructive pulmonary disease stage I/II (FEV1 ≥ 50%) ;
* Chronicle obstructive pulmonary disease stage III/IV (FEV1 < 50%) from may 2019 (ethical approvement granted)
* Weight ≤ 90kg ;
* Eligible for pulmonary rehabilitation.

Exclusion Criteria:

* Pregnant woman or likely to be ;
* Patient under guardianship ;
* Contraindication to cardiopulmonary exercise testing ;
* Patient medically treated with heart rate modulator (excluding oral B2-agonist) ;
* Patient treated with pacemaker or defibrillator ;
* History of lower limb impairment (i.e. peripheral artery disease, orthopedic disorder etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronicle obstructive pulmonary disease reffered for pulmonary rehabilitation.
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Relation between plateau heart rate (bpm) from the first and last 3 minutes of the 6-minute stepper test and heart rate (bpm) from first ventilatory threshold from cardiopulmonary exercise testing. | Heart rate (bpm) will be assessed during cardiopulmonary exercise testing with electrocardiogram. During the 2 6-minute stepper test, heart will be assessed with oximeter. All theses tests wil be carried out in a total time frame of 3 month maximum.
  Outcome (heart rate) during different tests will be continuously recorded. Relation will be adjusted for age and step count.

SECONDARY OUTCOMES:
Relation between minimal SpO2 (%)from the 6-minute stepper test and SpO2 (%) from first ventilatory threshold from cardiopulmonary exercise testing. | SpO2 will be assessed with oximeter. All theses tests wil be carried out in a total time frame of 3 month maximum.
  Outcome (SpO2 (%)) during different tests will be continuously recorded. Relation will be adjusted for age en step count.
Blood pressure (mmHg) before and after every 6-minute stepper test using electrical blood pressure device. | The outcome will be assessed before and after every 6-minute stepper test. The 2 6-minute stepper test will be carried out the same day (minimum 20 minute of rest between each test) for a total time frame of 1 day.
Steps during 6-minute stepper test using stepper device. | The 2 6-minute stepper test will be carried out on the same day (20 minute of rest between each test) for a total time frame of 1 day.

CONTACTS AND LOCATIONS:
Overall Officials: David Debeaumont, MD, Principal Investigator — CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de physiologie urinaire, digestive, respiratoire et sportive, Bois-Guillaume, France; Catherine Tardif, MD, Study Chair — CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de physiologie urinaire, digestive, respiratoire et sportive, Bois-Guillaume, France; Antoine Cuvelier, Prof, PhD, Study Chair — CHU-Hôpitaux de Rouen - Service de pneumologie, Hôpital de Bois-Guillaume, Rouen, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France.; Tristan Bonnevie, MsC, Study Chair — ADIR Association, Bois-Guillaume, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France; Francis-Edouard Gravier, PT, Study Chair — ADIR Association, Bois-Guillaume, France; Catherine Viacroze, MD, Study Chair — CHU-Hôpitaux de Rouen - Hôpital de Bois-Guillaume, Service de pneumologie, Bois-Guillaume, France; Jean-François Muir, Prof, PhD, Study Chair — CHU-Hôpitaux de Rouen - Service de pneumologie, Hôpital de Bois-Guillaume, Rouen, France ; UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France ; ADIR Association, Bois-Guillaume, France; Bouchra Lamia, Prof, PhD, Study Chair — UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France ; Service de pneumologie, Hôpital Jacques Monod 76290 Montivilliers; Jean Quieffin, MD, Study Chair — Service de pneumologie, Hôpital Jacques Monod 76290 Montivilliers; Guillaume Prieur, PT, MsC, Study Chair — Service de pneumologie, Hôpital Jacques Monod 76290 Montivilliers; Clément Médrinal, PT, MsC, Study Chair — UPRES EA 3830, Institut de Recherche et d'Innovation Biomédicale de Haute-Normandie, Université de Rouen, Rouen, France. Service de réanimation, Groupe Hospitalier du Havre, France; Pierre-Alexandre Hauss, MD, Study Chair — Service de pneumologie, Centre Hosptalier Intercommunal Elbeuf-Louviers-Val de Reuil
Locations (4):
- France (4):
  - ADIR Association, Bois-Guillaume
  - Centre Hostalier Intercommunal Elbeuf-Louviers-Val de Reuil, Elbeuf
  - Groupe Hospitalier du Havre, Le Havre
  - Centre Hospitalier de Morlaix, Morlaix

REFERENCES:
- [Derived] Bonnevie T, Clet A, Beaumont M, Smondack P, Combret Y, Medrinal C, Prieur G, Boujibar F, Muir JF, Cuvelier A, Grosbois JM, Debeaumont D, Artaud-Macari E, Gravier FE. Estimating endurance training intensity prescription from the 6-minute stepper test in people with chronic obstructive pulmonary disease - a multicenter cross-sectional study with external validation. Pulmonology. 2025 Dec 31;31(1):2486875. doi: 10.1080/25310429.2025.2486875. Epub 2025 Apr 11. PMID 40211884